CLINICAL TRIAL: NCT07384273
Title: Evaluating the Effectiveness of an Internet-based Therapy (iCARE) to Treat Symptoms of Postpartum Depression
Acronym: iCARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: University of Copenhagen (Other); Odense University Hospital (Other)
Responsible Party: Principal Investigator, Trine Munk-Olsen, Professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-0302-23; 23/15327 (Other: Region of Southern Denmark); 12.250 (Other: University of Southern Denmark); 514-1114/25-3000 (Other: Copenhagen University); 16-0302-23 (Other: The Danish Health Research Ethics Committee)
Record Dates: First submitted 2026-01-21; First posted 2026-02-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Postpartum Depression (PPD)
Keywords: Postpartum depression; Cognitive behavioural therapy; Internet-based therapy; Acceptance and commitment therapy; Randomised controlled trial
MeSH Terms: conditions — Depression, Postpartum | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Superiority, two-arm, randomised controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based therapy (iCARE) and treatment as usual (Experimental): The iCARE program is a self-guided iCBT intervention that also incorporates selected exercises and approaches from ACT. The iCARE program consists of four core modules and four optional modules. Together, these exercises aim to enhance psychological flexibility, reduce negative thinking, and promote well-being in daily life.
  The core modules focus on self-care and mindfulness (Module 1), identifying and reframing unrealistic expectations with self-compassion (Module 2), increasing positive experiences and countering self-critical thoughts (Module 3), and recognizing and challenging thinking traps (Module 4). The additional optional modules provide strategies for practicing being present, communicating needs and asking for support, bonding with the baby, and coping with scary thoughts.
  Interventions: Behavioral: Internet-based therapy (iCARE) and treatment as usual
- Treatment as usual (Active Comparator): In Denmark, there is large variation in the available prevention and treatment municipalities offers for women experiencing symptoms of PPD. Some municipalities offer specialized psychological support and support groups, while others provide only basic follow-up by health nurses. Women can also be referred to their general practitioner, who can provide free ongoing follow-up and prescribe antidepressant medication if needed. Alternatively, it is possible to be referred to a privately practicing psychologist, usually with some out-of-pocket cost.
  Interventions: Other: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Internet-based therapy (iCARE) and treatment as usual — The iCARE program is a self-guided iCBT intervention that also incorporates selected exercises and approaches from ACT. The iCARE program consists of four core modules and four optional modules. Together, these exercises aim to enhance psychological flexibility, reduce negative thinking, and promote well-being in daily life.
  The core modules focus on self-care and mindfulness (Module 1), identifying and reframing unrealistic expectations with self-compassion (Module 2), increasing positive experiences and countering self-critical thoughts (Module 3), and recognizing and challenging thinking traps (Module 4). The additional optional modules provide strategies for practicing being present, communicating needs and asking for support, bonding with the baby, and coping with scary thoughts.
  Arms: Internet-based therapy (iCARE) and treatment as usual
Other: Treatment as usual (TAU) — In Denmark, there is large variation in the available prevention and treatment municipalities offers for women experiencing symptoms of PPD. Some municipalities offer specialized psychological support and support groups, while others provide only basic follow-up by health nurses. Women can also be referred to their general practitioner, who can provide free ongoing follow-up and prescribe antidepressant medication if needed. Alternatively, it is possible to be referred to a privately practicing psychologist, usually with some out-of-pocket cost.
  Arms: Treatment as usual

SUMMARY:
Postpartum depression (PPD) is a common and serious condition affecting 9.5% of women in high-income countries, and around 8% in Denmark. It shares core features with major depression, including low mood, loss of interest, and impaired functioning. Untreated PPD can persist for months, negatively impacting maternal well-being, child development, and family dynamics. In Denmark, systematic screening using the Edinburgh Postnatal Depression Scale (EPDS) is standard practice, but access to PPD treatment varies widely across municipalities.

Cognitive behavioral therapy (CBT) is the most effective psychological intervention for perinatal depression, yet limited availability and long wait times create barriers to access to care. Internet-based CBT (iCBT) offers a scalable, cost-effective alternative that can be delivered flexibly at home. Evidence supports the efficacy of self-guided iCBT for depression, though challenges such as high dropout rates have been reported. International trials in Norway, Portugal, Iran, South Korea, and the US have shown promising results for iCBT in perinatal populations. Some recent iCBT based interventions have also incorporated elements of Acceptance and Commitment Therapy (ACT) - which emphasizes psychological flexibility via mindfulness-based acceptance and values-driven action-and have demonstrated efficacy in reducing postpartum depression symptoms. These kinds of interventions (either iCBT or iCBT + ACT) have not yet been tested and evaluated in Denmark.

This clinical trial aims to evaluate whether adding an iCBT intervention with elements from ACT (iCARE) to treatment as usual (TAU) is more effective than TAU alone in reducing depressive symptoms in mothers with symptoms of PPD.

Moreover, a qualitative process evaluation of the iCARE will explore implementation, acceptability, and mechanisms of impact. Its primary aim is to understand how participants experience the iCARE intervention and TAU, focusing on implementation fidelity, acceptability, and contextual influences. The secondary aim is to explore perceived mechanisms of change (e.g., cognitive, emotional, behavioral) and barriers/facilitators to engagement.

ELIGIBILITY:
Inclusion Criteria:

* Given birth within 6 months
* Edinburgh Postnatal Depression Scale (EPDS) score above 7
* ≥age 18
* Access to the internet

Exclusion Criteria:

* Do not understand Danish language,
* Substance abuse or dependence
* Alcohol abuse, defined by a weekly consumption of alcohol exceeding 10 units
* A diagnosis of schizophrenia, other psychotic disorders or in immediate need of psychiatric treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2026-02-01 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Symptoms of postpartum depression | Baseline At 2 months (primary endpoint) At 6 months (secondary endpoint)
  The Edinburgh Postnatal Depression Scale (EPDS) is a validated screening questionnaire that measures symptoms of postnatal depression, such as low mood, anxiety, and loss of enjoyment, over the past week. It helps identify mothers who may need further assessment or support but does not provide a diagnosis. The primary outcome is the between-group difference in change from baseline to 2-month follow-up in EPDS score (range 0-30; higher scores indicate more severe symptoms). A clinically meaningful response is defined as a ≥3-point reduction from baseline. Participants will be categorized as responders/non-responders, and proportions will be reported for each group.

SECONDARY OUTCOMES:
Symptoms of anxiety | Baseline At 2 months (primary endpoint) At 6 months (secondary endpoint)
  The Generalized Anxiety Disorder assessment (GAD-7) is a validated self-report questionnaire designed to assess symptoms of generalized anxiety disorder and overall anxiety severity. It consists of seven items scored from 0 (not at all) to 3 (nearly every day), producing a total score ranging from 0 to 21. Higher scores indicate greater anxiety symptoms. While the GAD-7 was originally developed to measure Generalized Anxiety Disorder, it has also been validated as a general measure of symptom severity of anxiety across different anxiety disorders in heterogeneous samples. In this trial, changes in GAD-7 scores from baseline to 2 and 6 months will indicate whether the intervention reduces anxiety symptoms.
Health-related disability and functioning | Baseline At 2 months (primary endpoint) At 6 months (secondary endpoint)
  World Health Organization Disability Assessment Schedule (WHODAS 2.0) is a generic, internationally validated tool for assessing health-related disability and functioning. The 12-item version used here provides a total score from 0 (no disability) to 48 (severe disability). It captures the broader impact of mental health symptoms on daily functioning and quality of life. Changes from baseline to 2 and 6 months will help determine whether iCARE improves overall functioning beyond symptom reduction.
Automatic negative thoughts/negative self-statements | At 2-months (primary endpoint)
  The Automatic Thoughts Questionnaire (ATQ) measures the frequency of automatic negative thoughts (negative self-statements). The shortened 8 item version will be used. It includes 8 items rated on a 5-point Likert scale, assessing thoughts such as self-criticism, hopelessness, and personal failure. Scores range from 0 (few negative thoughts) to 32 (frequent negative thoughts). Evaluating between-group differences in ATQ at 2 months follow-up will indicate whether the intervention effectively targets maladaptive thinking patterns.
Parental Stress | At 2-months (primary endpoint)
  The Danish Parental Stress Scale (DPSS) measures stress related to parenting responsibilities. It consists of 18 items rated on a 5-point scale, with total scores ranging from 18 (low stress) to 90 (high stress). Assessing DPSS at 2 months will help determine whether the intervention reduces stress associated with caring for an infant.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Unit of Child and Adolescent Psychiatry, Department of Clinical Research, University of Southern Denmark, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The individual de-identified participant data will be stored in (Open Patient data Explorative Network) and access might be available for affiliated researchers under data governance and approvals. The code will be available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, Analytic Code